CLINICAL TRIAL: NCT05624372
Title: Speech Perception in Noise in Children With ADHD
Acronym: ME
Status: Recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Maya Elazar, Principal Investigator, Sheba Medical Center
Other Study IDs: SHEBA-17-3855-ME-CTIL
Record Dates: First submitted 2018-05-21; First posted 2022-11-22 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: no Conditions
MeSH Terms: interventions — Hearing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Investigator: Child and Adolescent Psychiatrists, Speech Therapists
- Participant: Kids aged 4-18 diagnosed with ADHD
  Interventions: Diagnostic Test: hearing and cognitive assessment

INTERVENTIONS:
Diagnostic Test: hearing and cognitive assessment — psychiatric assessment, hearing assessment and brief cognitive assessment
  Groups: Participant

SUMMARY:
We are going to assess an ability of speech perception in voice in children diagnosed with ADHD (Attention Deficit Hyperactivity Disorder), comparing to normal control group. This is an attempt to understand the factors influencing on this ability.

DETAILED DESCRIPTION:
Participants will undergo a battery of hearing tests -Standard Hearing Test; Speech Perception in Noise - Hebrew Matrix; Transient Evoked Otoacoustic Emission (TEOAE) and cognitive tests - Working Memory Test (from (Wechsler Intelligence Scale for Children, WISC); Visual Attention Test (TMT (Trail Making Test)); Non-Verbal Intelligence Test (RAVEN)

ELIGIBILITY:
Inclusion Criteria:

* Research group: Kids diagnosed with ADHD, without previous hearing problems.
* Control group: Kids with regular development without previous hearing problems.

Exclusion Criteria:

For both groups:

* Having previous hearing problems or disorders
* Other psychiatric disorders
* Treatment with psychiatric medications other than stimulants
* Having autism
* Having severe learning disabilities.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Kids aged 4-18, diagnosed with ADHD, who get treatment and follow-ups in the ADHD outpatient clinic in the Sheba Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Speech perception in noise | 1 day
  Hebrew Matrix

CONTACTS AND LOCATIONS:
Locations (1):
- ADHD Medical Clinic, Child and Adolescent Psychiatry Unit, Sheba Medical Center, Ramat Gan, Israel